CLINICAL TRIAL: NCT02537847
Title: A Randomized Controlled Trial of Sitafloxacin and Ertapenem Treatment for Acute Pyelonephritis Caused by Extended-Spectrum ß-lactamase-producing Escherichia Coli
Brief Title: Sitafloxacin and Ertapenem Treatment for Acute Pyelonephritis Caused by Escherichia Coli
Acronym: SETAP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Chitprasong Malaisri, Ramathibodi Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sitafloxacin123
Record Dates: First submitted 2015-08-02; First posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Infection Due to Escherichia Coli; Acute Pyelonephritis
Keywords: Sitafloxacin; Extended-Spectrum ß-lactamase-producing Escherichia coli; Treatment for Acute Pyelonephritis; Ertapenem
MeSH Terms: conditions — Escherichia coli Infections | interventions — sitafloxacin; Fluoroquinolones; Ertapenem; Carbapenems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitafloxacin group (Experimental): The first third days of treatment was open label and all patients were given intravenous carbapenems. After day 3, the patients were randomized to either sitafloxacin group or ertapenem group by the use of a computer-generated random number allocation schedule and block size of four. The patients were allocated to the sitafloxacin group or ertapenem group using the sealed envelope method.
  Interventions: Drug: Sitafloxacin
- control group (Active Comparator): Intervention was prescribed ertapenem for patients.
  Interventions: Drug: Ertapenem

INTERVENTIONS:
Drug: Sitafloxacin — The patients in intervention group will receive carbapenem for the first 3 days then sitafloxacin for 7 days. Total of treatment duration is 10 days.
  Other Names: fluoroquinolone
  Arms: Sitafloxacin group
Drug: Ertapenem — Control group will be given ertapenem only for 10 days.
  Other Names: carbapenem
  Arms: control group

SUMMARY:
The aim of the investigators' study was to evaluate oral and non carbapenem antimicrobial agents which can be used in outpatient for the treatment of non-bacteremic acute pyelonephritis caused by Extended Spectrum Beta Lactamase Escherichia coli. This study was conducted to compare the clinical and bacteriological outcomes of patients with non-bacteremic acute pyelonephritis caused by Extended Spectrum Beta Lactamase Escherichia coli who were treated with intravenous (IV) carbapenems followed by oral sitafloxacin or IV ertapenem.

DETAILED DESCRIPTION:
A prospective randomized controlled trial of patients with a presumptive diagnosis of acute pyelonephritis caused by Extended Spectrum Beta Lactamase-producing pathogen was performed. Carbapenems was initially given to all patients. After day 3, patients were randomized to receive either oral sitafloxacin (100 mg twice daily) or intravenous ertapenem. The regular course of treatment was completed within 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Acute pyelonephritis by definition
* Positive urine culture for Extended Spectrum Beta Lactamase Escherichia coli ≥105 colony forming unit/mL
* Voluntarily consented to be enrolled in the study

Exclusion Criteria:

* Severe sepsis or septic shock
* Mixed organism of urine culture
* Positive blood culture
* Has other source of infection
* Has mechanical abnormality of urinary tract
* Immunocompromised conditions
* Retained Foley's catheter
* Pregnancy or lactation
* Previous urinary tract infections within 4 weeks
* Contraindicated for fluoroquinolones and carbapenems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-09 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
no symptoms of urinary tract infection | 30 days
  no fever, dysuria, back pain, nausea and vomiting

SECONDARY OUTCOMES:
no evidence of Extended Spectrum Beta Lactamase Escherichia coli in urine culture | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Sasisopin Kiertiburanakul, Study Director — Ramathibodi Hospital Mahidol University
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Bangkok, Bangkok, Thailand